CLINICAL TRIAL: NCT03229694
Title: Effect of Endothelin Receptor Blocker Tracleer on Toruniquet-associated Hypertension During Total Knee Arthroplasty
Brief Title: the Effect of Tracleer on Tourniquet-associated Hypertension
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuzhou Medical University (Other)
Responsible Party: Principal Investigator, Su Liu, Associtate professor, Xuzhou Medical University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: XYFY-2017-068
Record Dates: First submitted 2017-07-20; First posted 2017-07-25 (Actual); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Tourniquets; Hypertension; Bosentan
MeSH Terms: conditions — Hypertension | interventions — Bosentan; Tablets; Endothelin Receptor Antagonists

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Tracleer (or Bosentan) (Experimental): Tracleer (Tracleer 125Mg Tablet) was administered orally at two hours before surgery and six hours after surgery
  Interventions: Drug: Tracleer 125Mg Tablet
- Placebo (Placebo Comparator): Placebo was administered orally at two hours before surgery and six hours after surgery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tracleer 125Mg Tablet — Tracleer was administered orally at two hours before surgery and six hours after surgery.
  Other Names: Bosentan; endothelin receptor antagonist
  Arms: Tracleer (or Bosentan)
Drug: Placebo — Placebo was administered orally at two hour before surgery and six hours after surgery.
  Arms: Placebo

SUMMARY:
Tourniquet is widely used in orthopedic surgery. However, prolonged tourniquet inflation may cause a gradual rise in blood pressure, which named as tourniquet-associated hypertension. Thus, to effectively prevent the tourniquet related hemodynamic responses is important for patients receiving limb surgery.

Tracleer is an endothelin receptor antagonist indicated for the treatment of pulmonary arterial hypertension. Tracleer can also be used to treat retistant hypertension. At present trial, the investigators are going to investigate the effect of Tracleer on tourniquet-associated hypertension during total knee arthroplasty.

DETAILED DESCRIPTION:
At present study, the investigators will use endothelin receptor antagonist, Tracleer (Bosentan), to investigate the effect of Tracleer on tourniquet-associated hypertension during unilateral total knee arthroplasty, and evaluate its safety and effectivity. The purpose of this study is to find a new therapy to prevent and treat tourniquet-associated hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Patients underwent selected total knee arthroplasty under general anesthesia
* ASA II-III
* 18~65 years old
* Signed informed consent voluntarily

Exclusion Criteria:

* Do not apply tourniquet during the surgery
* Patients underwent emergency surgery
* Having applied tourniquet in last three months
* Patients underwent bilateral total knee arthroplasty
* Dysfunction of liver or kidney
* Anemia (Hb <90 g/L)
* Serious myocardial disease (eg. coronary heart disease, heart failure, severe arrhythmia)
* Coagulation disorder
* Diabetic
* Leukocyte higher than normal value
* Pneumonia, asthma, chronic obstructive pulmonary disease
* Hypotension before surgery (systolic pressure < 90 mmHg)
* Pregnant woman or puerpera
* Having being enrolled in other clinical trial in last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2017-08-01 (Estimated); Primary Completion 2018-04-01 (Estimated); Study Completion 2018-05-01 (Estimated)

PRIMARY OUTCOMES:
Maximum rate of change in systolic blood pressure (MR) | 24 hours after surgery
  During the observation, MR=(the highest value of systolic blood pressure - the baseline of systolic pressure ) / the baseline of systolic pressure

SECONDARY OUTCOMES:
the concentration of endothelin-1, 5-hydroxytrypatamine, and norepinephrine | baseline and intraoperative
  test the concentration of endothelin-1, 5-hydroxytrypatamine, and norepinephrine in plasma at different time point
visual analog scale | 24 hrs after surgery
  assess the efficacy of analgesia using visual analog scale (VAS)

CONTACTS AND LOCATIONS:
Overall Officials: Su Liu, doctor, Principal Investigator — The Affiliated Hospital of Xuzhou Medical University
Locations (1):
- The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided